CLINICAL TRIAL: NCT00006268
Title: Interstitial Infusion of IL 13-PE38QQR Cytotoxin in Recurrent Malignant Glioma: Phase I/II Study
Brief Title: Immunotoxin Therapy in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Approaches to Brain Tumor Therapy Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068211; NABTT-9903; JHOC-NABTT-9903; NEOPHARM-TS-G1-TI4; NEOPHARM-IL13PEI-001-R03
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Glioma; Gliosarcoma | interventions — IL13-PE38

INTERVENTIONS:
Biological: cintredekin besudotox
Drug: isolated perfusion
Procedure: conventional surgery

SUMMARY:
RATIONALE: Immunotoxins can locate tumor cells and kill them without harming normal cells. This may be an effective treatment for malignant glioma.

PURPOSE: Phase I/II trial to study the effectiveness of immunotoxin therapy in treating patients who have malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects and maximum tolerated dose (MTD) of interstitial interleukin-13 PE38QQR immunotoxin in patients with malignant glioma.
* Determine the response rate, duration of response, time to response, overall survival, and time to progression in patients treated with this regimen.
* Determine the toxic effects of this drug at the MTD in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients undergo stereotactic biopsy of brain tumor followed by CT guided stereotactic placement of 2 intratumoral catheters on day 0. Patients with histologically confirmed malignant glioma receive interleukin-13 PE38QQR immunotoxin interstitially over 96 hours beginning on day 1. Patients with a residual enhancing mass undergo repeat catheter placement on day 56 and then receive a second interstitial infusion beginning on day 57 in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of interleukin-13 PE38QQR immunotoxin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6 patients experience dose-limiting toxicity. Additional patients are treated at the MTD.

Patients are followed every 8 weeks.

PROJECTED ACCRUAL: A maximum of 30 patients will be accrued for phase I of the study within 6 months and a total of 12-35 patients will be accrued for phase II of the study within 10-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven malignant glioma (grade 3 or 4)

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Malignant mixed oligoastrocytoma
* Must have undergone cranial radiotherapy with tumor dose of at least 48 Gy and at least 12 weeks prior to study
* Must have undergone supratentorial brain tumor surgery or biopsy
* Must have radiographic evidence of recurrent or progressive supratentorial tumor compared with prior study

  * Must have solid portion measuring 1.0-5.0 cm in maximum diameter
  * Maximum of 1 satellite lesion allowed if separated from the primary mass by less than 3 cm
  * No tumor crossing the midline
  * No leptomeningeal tumor dissemination
  * No impending herniation or spinal cord compression
* No uncontrolled seizures

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Hemoglobin at least 10 g/dL
* Platelet count at least 100,000/mm^3

Hepatic:

* PT and PTT no greater than upper limit of normal (ULN)
* SGOT and SGPT no greater than 2.5 times ULN
* Bilirubin no greater than 2.0 mg/dL

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior intralesional chemotherapy for malignant glioma
* At least 3 weeks since other prior chemotherapy (6 weeks since prior nitrosoureas) and recovered
* No concurrent chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed, but dose must remain stable or be tapered during study

Radiotherapy:

* See Disease Characteristics
* No prior focal radiotherapy (e.g., any form of stereotactic radiotherapy or brachytherapy) for malignant glioma

Surgery:

* See Disease Characteristics

Other:

* Recovered from any prior therapy
* No other concurrent investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Weingart, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (11):
- United States (11):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - National Institute of Neurological Disorders and Stroke, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas